CLINICAL TRIAL: NCT01050920
Title: Study of Genetic Factors Other Than CYP2C9 and VKORC1 That Influence Warfarin Dose Requirements in a South-east Asian Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: PK03/32/09
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Blood Collection
  Interventions: Biological: Blood collection

INTERVENTIONS:
Biological: Blood collection

SUMMARY:
Warfarin is a commonly used anti-coagulant, but has a narrow therapeutic index and wide inter-individual and inter-ethnic variation in dose requirements. Several genetic and non-genetic factors have been identified that could influence warfarin dose requirements. However, current known predictive factors could only explain about 50-60% of warfarin dose variability. Inter-ethnic differences in genetic influences on warfarin dose requirements also exist. We hypothesize that genetic factors other than CYP2C9 and VKORC1 may influence warfarin dosing and serve to further optimize warfarin dosing.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving maintenance warfarin therapy with a stable therapeutic international normalized ratio (INR) between 2 and 3 for at least 3 months,
* patients recruited from the anticoagulation clinics at the National University Hospital and Tan Tock Seng Hospital in Singapore between June 2002 and June 2004 for a previous genotyping study (C/00/510, NUH; C/00/535, TTSH, PI-Dr Goh Boon Cher).

Exclusion Criteria:

* patients below 21 years old, or
* patients with liver disease, malabsorption or chronic diarrheal diseases, or
* patients taking drugs that may potentially interact with warfarin.

Dietary advice to avoid foods that may interfere with warfarin pharmacokinetics will be given to patients during warfarin therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Germline DNA will be genotyped for variants in genes in the anti-coagulation pathway, including CYP4F2, GGCX and EPHX1. The germline DNA was previously collected from a warfarin study (C/00/510, NUH, C/00/535, TTSH, PI-Dr Goh Boon Cher). Samples were anonymized, and data analysis will be done without patient identifiers. Germline DNA previously collected from 279 patients who were on maintenance warfarin dose will be genotyped.
  The clinical data that has been collected and will be used for the study include: gender, race, age, body weight, maintenance warfarin dose, serum albumin, two consecutive stable INR values, and indications for warfarin use.
Sampling Method: Probability Sample
Dates: Start 2013-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To identify genetic variants other than CYP2C9 and VKORC1 that may influence warfarin dose requirements in a multi-ethnic population in Singapore.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Hirsh J, Fuster V, Ansell J, Halperin JL; American Heart Association/American College of Cardiology Foundation. American Heart Association/American College of Cardiology Foundation guide to warfarin therapy. J Am Coll Cardiol. 2003 May 7;41(9):1633-52. doi: 10.1016/s0735-1097(03)00416-9. No abstract available. PMID 12742309
- [Background] Poller L, Taberner DA. Dosage and control of oral anticoagulants: an international collaborative survey. Br J Haematol. 1982 Jul;51(3):479-85. doi: 10.1111/j.1365-2141.1982.tb02805.x. PMID 7104231